CLINICAL TRIAL: NCT06635330
Title: A Phase I/II Single Arm Study, Safety and Efficacy Assessment of the CD19 CAR T Cell on Pediatric Patients with Relapsing or Refractory B Cell Acute Lymphoblastic Leukemia (r/r B-ALL)
Brief Title: Safety and Efficacy of CAR T Cell Therapy in Patients with R/r B-ALL
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kara Yakhteh Tajhiz Azma Company (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IR.NREC.1403.003
Record Dates: First submitted 2024-10-01; First posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Relapse/Refractory B-cell Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Recurrence; Burkitt Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Anti-CD19 CAR-T treatment group (Experimental)
  Interventions: Biological: anti-CD19 CAR T cell therapy

INTERVENTIONS:
Biological: anti-CD19 CAR T cell therapy — Anti-CD19 CAR-T cell therapy for R/R B-ALL pediatric patients. For patients 50 kg and less: 0.2 to 5 in ten to the power of six live CAR+ T cells per kilogram of body weight/ For patients over 50 kg: 0.1 to 2.5 in ten to the power of eight live CAR+ T cells (without considering weight).

SUMMARY:
The goal of this clinical trial is to evaluate the safety and efficacy of CD19 CAR-T cells in pediatric patients of all genders, aged 2 to 18 years, with relapsing or refractory B cell acute lymphoblastic leukemia (r/r B-ALL). The main questions it aims to answer are as following:

1. What is the percentage of patients with overall remission rate (ORR) of complete response (CR) or complete remission with incomplete blood count recovery (CRi)?
2. What is the rate of Event-free survival at first month and 2-3 months after intervention?
3. What is the rate of Overall survival at first month and at 3 months after the intervention?

DETAILED DESCRIPTION:
B-cell acute lymphoblastic leukemia (B-ALL), as the most common type of pediatric tumor, is identified by unregulated cell proliferation of immature lymphoid cells that can infiltrate the bone marrow and blood. Also, relapse and refractory B-ALL (R/R B-ALL) is the main reason of global mortality due to the constraints of combination chemotherapy.

Over the past few years, substantial advancements have been made in treatment of ALL, specifically in the R/R context. Chimeric antigen receptor T (CAR-T) cells are a type of cancer immunotherapy treatment that function through modification of patient T cells to express CAR antigen on their surface. CAR-T cells aimed at CD19 have demonstrated promising activity in treatment of r/r B-ALL. In this study we aim to evaluate safety and efficacy of Anti-CD19 CAR T cell therapy in children with R/R B-ALL.

ELIGIBILITY:
Inclusion Criteria:

* Ages 2 to 18 years with relapsed or refractory CD19+ B-ALL
* Presence of disease in the bone marrow
* Able to tolerate the apheresis process
* Life expectancy > 12 weeks
* Lansky or Karnofsky score > 50%
* At least 7 days passed since the last chemotherapy and the last treatment with corticosteroids
* Informed consent
* Having potential donor for stem cell transplantation

Exclusion Criteria:

* Presence of active malignancy other than the disease under study
* Chloroma and leukemic infiltration on MRI or significant neurological symptoms
* Any CNS disorder
* Presence of active GVHD
* Radiation therapy within last 14 days
* History of Anti-CD19 or Anti-CD20 therapy
* Donor lymphocyte injection or other cell therapy methods within the last 30 days
* Presence of severe active infection
* Organ dysfunction

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2026-09-22 (Estimated); Study Completion 2027-09-22 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with overall remission rate (ORR) of complete response (CR) or complete remission with incomplete blood count recovery (CRi) | First month and 2-3 months after intervention
Overall survival | First month and 3 months after intervention
Incidence of cytokine release syndrome: grade 3 and 4 | First month and 3 months after intervention
Incidence of Immune effector cell-associated neurotoxicity syndrome (ICANS): grade 3 and 4 | First month and 3 months after intervention
Event-free survival | First month and 2-3 months after intervention

SECONDARY OUTCOMES:
Percentage of patients with overall remission rate (ORR) of complete response (CR) or complete remission with incomplete blood count recovery (CRi) | 6 months and 12 months after intervention
Investigation of Minimal residual disease in patient | First month and 2-3 months after intervention
Incidence of cytokine release syndrome: grade 3 and 4 | 6 months and 12 months after intervention
Incidence of Immune effector cell-associated neurotoxicity syndrome (ICANS): grade 3 and 4 | 6 months and 12 months after intervention
Incidence of tumor lysis syndrome (TLS) | Months 1, 3, 6, and 12 after the intervention
Incidence of leukopenia | Months 1, 3, 6, and 12 after the intervention
Incidence of infection | Months 1, 3, 6, and 12 after the intervention
Event-free survival | 6 months and 12 months after intervention
Overall survival | 6 months and 12 months after intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric cell and gene therapy research center, Children medical center, Tehran, Tehran Province, Iran